CLINICAL TRIAL: NCT05644574
Title: Posterior Surgical Management of Post-Traumatic Kyphosis
Brief Title: Surgical Management of Post-Traumatic Kyphosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haytham AlmEdden Ahmad, principle investigator, Assiut University
Other Study IDs: Surgery in PTK
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Post-Traumatic Kyphosis
Keywords: Post-Traumatic Kyphosis; Posterior only surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to examine the safety and efficacy of posterior sugary only in addressing post traumatic kyphosis. The main question[s]it aims to answer are:

Is it a safe procedure? Is it a sufficient approach to address deformity? Participants will be managed by posterior only surgery to address their deformity and will be assessed for the radiological and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

- All patients with age range from 18-65 years old with PTK underwent corrective surgery and have been followed for at least 2 years with complete documentation.

Exclusion Criteria:

* Traumatic cervical spine deformities
* Pathologic fracture spine
* Congenital or developmental cases
* Degenerative cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with age range from 18-65 years old with PTK underwent posterior only corrective surgery and have been followed for at least 2 years with complete documentation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
change in degree of kyphosis | 2 years
  we will measure the kyphosis in pre operative radiogragh and post operative radiograph to detect the change in the degree and the correction achieved after posterior only operative correction